CLINICAL TRIAL: NCT04882787
Title: Validation of 2 Novel BTE Hearing Aid Models Varying With Respect to Regular-power or Super-power Gain Specifications
Brief Title: Validation of Novel BTE and SP Hearing Aid Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Sonova Canada Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 378
Record Dates: First submitted 2021-05-04; First posted 2021-05-12 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2023-06

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: 2 groups based on hearing aid gain needs; one similar intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BTE hearing aid model (Experimental): BTE or SP-BTE (super power) hearing aid fitting
  Interventions: Device: BTE hearing aid

INTERVENTIONS:
Device: BTE hearing aid — Amplification

SUMMARY:
Participants will wear one set of 2 different BTE hearing aid models based on the gain required by their hearing loss. The hearing aids will be programmed based on a prescriptive approach and participants will be sent out for either one home trial with the less powerful BTEs or for two home trials with the SP (super power) BTEs.

DETAILED DESCRIPTION:
During this study each participant will be asked to wear a set of BTE hearing aids home and wear them daily. We will be assessing their evaluation of the BTEs during and after their home field trial. They will be asked to report on their use with different apps/accessories. Subjective performance ratings will be collected.

ELIGIBILITY:
Inclusion Criteria:

* hearing aid candidacy (N2-N7 hearing loss)
* healthy outer and middle ears
* ability to complete questionnaires
* willingness to use smartphone
* informed consent documented by a signature
* willingness to wear a binaural BTE fitting
* willingness to use app and accessories
* willingness to adhere to COVID protocols

Exclusion Criteria:

* contraindications to the MD in this study: known hypersensitivity or allergy to investigational product/earmold
* limited mobility/not able to attend appointments
* limited ability to describe listening impressions/experiences
* inability to produce a reliable hearing test result
* limited dexterity - to point that participant cannot manage hearing aid insertion/removal
* known psychological disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinyu Qian, PhD, Principal Investigator — Sonova AG
Locations (1):
- Unitron Hearing, Kitchener, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gabrielsson A, Schenkman BN, Hagerman B. The effects of different frequency responses on sound quality judgments and speech intelligibility. J Speech Hear Res. 1988 Jun;31(2):166-77. doi: 10.1044/jshr.3102.166. PMID 3398490
- [Background] Valente M, Van Vliet D. The Independent Hearing Aid Fitting Forum (IHAFF) Protocol. Trends Amplif. 1997 Mar;2(1):6-35. doi: 10.1177/108471389700200102. No abstract available. PMID 25425874
- [Background] Likert, Rensis. A technique for the measurement of attitudes. Archives of Psychology. 1932; 140: 1-55.

RESULTS

PARTICIPANT FLOW:
Groups:
- BTE Hearing Aid Model: (same arm, different group) hearing aid providing 'less' amplification for less severe hearing losses (mild to moderately-severe) BTE hearing aid: Amplification
- SP-BTE (Super Power) Hearing Aid Model: (same arm, different group) hearing aid providing more amplification for greater (severe to profound) hearing losses BTE hearing aid: Amplification
Period: Overall Study
Arm/Group | BTE Hearing Aid Model | SP-BTE (Super Power) Hearing Aid Model
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: mild to moderately-severe hearing loss appropriate for 'regular' BTE fitting with 3 week take home trial vs severe to profound hearing loss appropriate for 'super power' BTE fitting with 7 week take home trial duration
Groups:
- BTE Hearing Aid Model: BTE hearing aid fitting
  BTE hearing aid: Amplification
- SP-BTE Hearing Aid Model: Super power BTE hearing aid fitting
  BTE hearing aid: Amplification
- Total: Total of all reporting groups
Arm/Group | BTE Hearing Aid Model | SP-BTE Hearing Aid Model | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 5 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 7 | 7 | 14
Hearing aid candidate [Count of Participants; unit: Participants] | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 'Total Impression' Sound Quality as 'Good'
Description: Participants with 'good' response of 7 or higher on 'Total Impression' scale; Gabrielsson citation/article includes seven perceptual scales and a scale for 'Total Impression' which is described as 'an overall judgment of how good you think the reproduction is'.
  Possible scores from 0 to 10 with descriptors provided: 0 (min), 1 (very bad), 3 (rather bad), 5 (midway), 7 (rather good), 9 (very good), 10 (max) A higher score reflects a better outcome.
Time Frame: final appointment (end of 3 weeks home trial for BTE model, end of 7 weeks home trial for SP-BTE model)
Population: Participant (fit with hearing aids binaurally)
Measure: Count of Participants; unit: Participants
Groups:
- SP-BTE Hearing Aid Model: super power hearing aid fitting BTE hearing aid: Amplification
Arm/Group | BTE Hearing Aid Model | SP-BTE Hearing Aid Model
Number analyzed (Participants) | 7 | 7
Participants
  Count of participants who reported score of 7 or above | 7 | 6
  Count of participants who reported score of 6 or below | 0 | 1

2. Secondary Outcome: Number and Percentage of Participants Reporting No Reboots
Description: Participants to report perceived unwanted reboots of the hearing aids as an indicator of system stability (with use of 2.4 GHz connectivity including accessories and smartphones). Possible responses for perceived reboots (i.e., instances when the amplified sound dropped out and then returned) are: 'No (0) reboots perceived' or 'Reboots perceived (1 or more)'.
Time Frame: at any time during home trial, reported at or by final appointment(end of 3 weeks home trial for BTE model, end of 7 weeks home trial for SP-BTE model)
Population: Participant (wearing binaural amplification, using accessories and smartphones with 2.4 GHz connectivity)
Measure: Count of Participants; unit: Participants
Groups:
- SP BTE Hearing Aid Model: super power hearing aid fitting
Arm/Group | BTE Hearing Aid Model | SP BTE Hearing Aid Model
Number analyzed (Participants) | 7 | 7
Participants
  Count of participants reporting 0 reboots | 6 | 6
  Count of participants reporting 1 or more reboots | 1 | 1

3. Secondary Outcome: Number of Participants Reporting Perceived Differences With Both of the App Boost Controls
Description: Number of SP-BTE participants reporting perceived differences from adjustment of the app's Boost controls.
  Stimuli were presented in a sound room to check the Clarity & Comfort Boosts in the app (available in Automatic Program). To comment on the effect of the Boosts, participants listened to simulated acoustic scenarios, initially under default settings (i.e., with no Boost), then with each Boost (Comfort then Clarity) activated separately (by pressing a button on a screen in the app).
  Yes/No answer to confirm a perceived difference -- 'Did you notice a difference?'
Time Frame: initial appointment (day of fitting of hearing aids)
Population: SP-BTE Participant (wearing binaural amplification, using smartphone app interactive controls); no data were collected for participants in the "BTE hearing aid model" Arm/Group.
Measure: Count of Participants; unit: Participants
Arm/Group | SP-BTE Hearing Aid Model
Number analyzed (Participants) | 7
Participants
  Count of participants reporting a perceived difference, i.e. "yes" with both of the Boost controls | 7
  Count of participants reporting no perceived difference, i.e. "no" with both of the Boost controls | 0

4. Secondary Outcome: Number of Participants Reporting Perceived Differences With Both of the App Slider Controls
Description: Number of SP-BTE participants reporting perceived differences from adjustment of two of the app's Slider controls.
  Stimuli were presented in a sound room to check the Enhance Speech and Reduce Noise sliders in the app (available in Manual Program). To comment on the effect of the Sliders, participants were asked to adjust the Enhance Speech and Reduce Noise Sliders (separately) to the Maximum and Minimum settings (by sliding the setting indicator across the available range).
  Yes/No answer to confirm a perceived difference -- 'Did you notice a difference?'
Time Frame: initial appointment (day of fitting of hearing aids)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SP-BTE Hearing Aid Model
Number analyzed (Participants) | 7
Participants
  Count of participants reporting a perceived difference, i.e. "yes" with both of the Slider controls | 6
  Count of participants reporting no perceived difference, i.e. "no" with both of the Slider controls | 1

ADVERSE EVENTS:
Time Frame: 2 months
Description: Point of Care Risk Assessment conducted at each visit, including questions regarding health primarily due to COVID (in addition to online COVID screening form) e.g., how are you feeling? and ensuing discussion
Groups:
- SP-BTE Hearing Aid Model: SP-BTE (super power) hearing aid fitting
  BTE hearing aid: Amplification
Arm/Group | BTE Hearing Aid Model | SP-BTE Hearing Aid Model
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT04882787/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT04882787/ICF_001.pdf